CLINICAL TRIAL: NCT06287411
Title: Role of FAPI PET/MR Combined With Gadoxetate Disodium in Assessing Hepatic Malignancies
Status: Recruiting | Type: Observational
Sponsor: Xiao Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 202436
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Malignancies
Keywords: hepatic malignancies; FAPI; PET/MR; gadoxetate disodium; FDG

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — histopathological findings obtained from biopsy or resected surgical specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FAPI PET/MR combined with gadoxetate disodium — Patients with clinical suspected hepatic malignancies will receive the FAPI PET/MR.

SUMMARY:
This study aimed to prospectively evaluate the utility of fibroblast activation protein inhibitor (FAPI) positron emission tomography (PET)/magnetic resonance (MR) combined with gadoxetate disodium in patients with clinical suspected hepatic malignancies (lesion diameter ≤ 3.0cm), with histopathological findings obtained from biopsy or resected surgical specimens, or follow-up results as reference standards.

DETAILED DESCRIPTION:
1. Clinical and biological data, including the course of disease, underlying liver disease (hepatitis or cirrhosis), serum alpha-fetoprotein, carcinoembryonic antigen and carbohydrate antigen 19-9 levels were collected from each patient.
2. PET image analysis: Each patient underwent both FAPI and fluorodeoxyglucose (FDG) PET/MR, including T1-weighted imaging (T1WI), T2-weighted imaging (T2WI), diffusion-weighted imaging (DWI), apparent diffusion coefficient (ADC) and gadoxetate disodium-enhanced MRI. Record and evaluate the following indicators: the maximum standardized uptake value (SUVmax) of lesions, the target-to-background ratio (TBR) which was calculated by dividing the SUVmax of the lesion by the background SUVmean obtained from nontumor liver tissue.
3. Pathological analysis: Hematoxylin and eosin staining and immunohistochemical analyses will be performed. Immunohistochemical analysis will be used to investigate the expression of glucose transporter-1 (GLUT-1) and fibroblast activation protein (FAP).

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years of age at the time of consent;
2. Patients with suspected, newly diagnosed, or previously treated liver cancer;
3. Estimated creatinine clearance > 30ml/min;
4. Provided written informed consent authorisation before participating in the study.

Exclusion Criteria:

1. Allergic to the gadoxetate disodium；
2. MRI contraindications, not limited to cardiac implantable electronic devices and claustrophobia;
3. Weight > 90Kg;
4. Pregnancy or lactation;
5. Active inflammation may affect FAPI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects the investigators selected are adults who are not restricted by gender.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 2 years
  sensitivity, specificity, accuracy, positive and negative predictive values

SECONDARY OUTCOMES:
Quantitative parameters of PET/MR | completed within one week after the PET examination
  the maximum standardized uptake value and tumour-to-background ratios

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, Ph.D, Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo W, Pang Y, Yao L, Zhao L, Fan C, Ke J, Guo P, Hao B, Fu H, Xie C, Lin Q, Wu H, Sun L, Chen H. Imaging fibroblast activation protein in liver cancer: a single-center post hoc retrospective analysis to compare [68Ga]Ga-FAPI-04 PET/CT versus MRI and [18F]-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1604-1617. doi: 10.1007/s00259-020-05095-0. Epub 2020 Nov 11. PMID 33179149